CLINICAL TRIAL: NCT05477784
Title: Enhancing Connections-Palliative Care: A Cancer Parenting Program for Patients With Advanced Cancer and Their Children
Brief Title: Cancer Parenting Program for the Enhancement of the Quality of Life of Patients With Advanced Cancer and Their Children
Acronym: EC-PC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment rates to the trial were lower than projected and anticipated.
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RG1122669; R01NR019987-01A1 (NIH); STUDY00011221 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2022-08714 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Parenting; Parent-Child Relations; Cancer; Survivorship; Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Intervention Model Description: 2-group randomized control trial: experimental and alternative treatment control group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only biostatistician will be unmasked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (enhancing connections-palliative care program) (Experimental): Patients receive the 5-session EC-PC program bi-weekly with a patient educator about ways to help them talk to and support their child.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Group II (educational material) (Active Comparator): Patients receive carefully selected educational booklet that discuss ways to talk about their cancer with their child and a scripted phone call from a trained phone counselor on study.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive EC-PC program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education
  Arms: Group I (enhancing connections-palliative care program)
Other: Informational Intervention — Receive education booklet
  Arms: Group II (educational material)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial examines the usefulness of two educational programs for parents with late-stage cancer who have a 5 - 17 year old child. The programs are designed to enhance the quality of the parent-child relationship and add to the parent's confidence in managing the impact of their cancer on their child. Educational programs may reduce anxiety and depression and improve the well-being and quality of life of parents with advanced cancers and their children.

Recruitment occurs nationally via referral to the Fred Hutch/University of Washington Cancer Consortium team.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (ENHANCING CONNECTIONS-PALLIATIVE CARE [EC-PC] PROGRAM): Patients receive the 5-session EC-PC program bi-weekly with a patient educator about ways to help them talk to and support their child.

GROUP II (CONTROL): Patients receive carefully selected educational booklet that discuss ways to talk about their cancer with their child and a scripted phone call from a trained phone counselor on study.

ELIGIBILITY:
Inclusion Criteria:

* Parents with any type of late-stage, non-curable cancer (determined by TNM stage IV cancer for solid tumors or 2 or more cycles of treatment failure with disease relapse in non-solid tumors)
* All therapies are allowable
* 23 years (yr.) to 68 yr. Age restriction exists for the patient based on parent having a child ages 5-17
* Patient must have a child (5yr. -17 yr.) living in the home at least 50% of the time and residential with non-ill parent or parent surrogate
* Read and write English as one of their languages of choice
* Have access to a telephone
* Ability to understand and the willingness to sign a written informed consent document. Read and write English as one of their languages of choice

Exclusion Criteria:

* Patient is in hospice at time of enrollment
* Non-ill co-parent does not consent to join study

Ages: 23 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy assessed by parents' mood (CES-D) | At 3 months post-baseline
  Depressed mood will be measured by the 20-item Center for Epidemiological Studies- Depression Scale (CES-D) (Benazon & Coyne, 2000; Lewis, Fletcher, Cochrane, & Fann, 2008; Radloff, 1977). The CES-D Scale measures the recent occurrence of symptoms of depression. For each symptom, the respondent indicates the frequency with which that symptom has occurred during the past week, from "rarely or none of the time (less than 1 day)" to "most or all of the time (5-7 days)." This measure has been well- accepted in both ill and non-ill samples. Internal consistency in three samples from the general population has been reported by Radloff (Radloff, 1977) and ranged between .84 to .85. Validity has been well- established, including its link to the broader concept of "distress" in cancer-related research (Benazon & Coyne, 2000; Coyne et al., 1987; Given et al., 2004) The internal consistency reliability is 0.85 or higher (Benazon & Coyne, 2000; Coyne et al., 1987; Given et al., 2004).
Treatment efficacy assessed by parents' anxiety [Spielberger State-Trait Anxiety (STAI, state scale)] | At 3 months post-baseline
  State anxiety will be measured by the state component of the State-Trait Anxiety Inventory. This 20-item self-report questionnaire evaluates current feelings of apprehension, tension, nervousness, and worry. The respondent circles a response that best depicts their current feelings best. Response options range from [1 - Not at all] to [5 - Very much so]. Sample items include "I feel calm", I am tense." Higher scores denote greater anxiety. Internal consistency reliability is 0.90 or above in community and population samples [Edwards and Clarke, 2004]
Parent's confidence in being able to talk with her child about the child's cancer-related concerns (CASE Help Child Subscale) | At 3 months post-baseline
  Parenting Self-efficacy: Measured by the Help Child subscale of the parent-reported cancer Self-efficacy Scale (CASE). The Help Child subscale (9 items) measures the parent's confidence in being able to talk with her child about the child's cancer-related concerns; e.g., "I can assist my child to talk out his/her worries about my cancer." Structured response options range from "Not at all confident" (1) to "Very confident." The internal consistency reliability The internal consistency reliabilities in the EC seminal trial with parents with early stage cancer was 0.97.
Parents' skills in helping their child cope and manage the toll of the parents' cancer (Connecting and Coping Subscale) | At 3 months post-baseline
  Parenting skills will be measured by the parent reported Parenting Skills Checklist: Connecting and Coping subscale developed by the study team and tested for reliability and validity in a 6-state randomized control trial (Lewis et al., 2015). The measure describes the observable interactional behaviors parents can use to assist their child disclose, discuss, and cope with the parent's cancer. The developmental-contextual model of parenting was the conceptual basis for the measure. An example item on the Connecting and Coping subscale includes, "I work with my child to help my child manage the child's stress related to my cancer."
Child-Behavioral Emotional Functioning: Anxious/Depressed, Internalizing, Externalizing scores on CBCL | At 3 months post-baseline
  The child's behavioral-emotional adjustment will be measured by the Anxious/Depressed, Internalizing and Externalizing scores of the CBCL which is part of the Child Behavior Checklist. This measure will be obtained from both the ill parent and the non-ill parent/parent surrogate. Response options range from 0 to 2 from "Not True (as far as you know)" to "Somewhat or Sometimes True" to "Very True or Often True." This score is part of the Internalizing score of the CBCL that measures the child's fearful, inhibited, and over-controlled behavior. The internal consistency reliabilities for the EC clinical trial were 0.90 for the Internalizing score and 0.94 for the Externalizing score. For the current study, we will use the CBCL form for 6-18 year-olds and its computer software.

SECONDARY OUTCOMES:
Effects of parents' symptom burden on treatment outcomes: Condensed Memorial Symptom Assessment scale (CMSAS) - Physiological symptoms subscale | At 3-months post-baseline
  Using Linear Mixed Models, will examine the moderator effects of the diagnosed parent's symptom burden on intervention outcomes. Will be assessed using the physiological symptoms subscale (range of scores 0-4).

CONTACTS AND LOCATIONS:
Overall Officials: Frances M Lewis, RN, MN, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Secondary analysis of data will be permitted after a specific plan is submitted to the Principal Investigator and Co-Investigators approve.
  Plan should make explicit the analysis sample, rationale for study, aims of secondary analysis, proposed data analysis to be used, timeline for completion of analysis, and agreement to cite the parent study with appropriate acknowledgment.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after filing FINAL Report to NINR, NIH and after the efficacy results and analysis of study aims are published.
Access Criteria: Scientists prepared with a PhD or equivalent degree will be granted access for secondary analysis, after their specific proposed plan is submitted and reviewed by PI and Co-Invesigators.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT05477784/ICF_000.pdf